CLINICAL TRIAL: NCT05719688
Title: Prospective, Multicenter, Randomized, Parallel Controlled Study to Evaluate the Safety and Efficacy of Thrombectomy System in the Intravascular Treatment of Acute Ischemic Stroke
Brief Title: Evaluate the Safety and Efficacy of Thrombectomy System in the Intravascular Treatment of Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Hengruihongyuan Medical Technology Co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRD01
Record Dates: First submitted 2022-11-20; First posted 2023-02-09 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mechanical thrombectomy:Thrombectomy system (Experimental): Subjects will be treated with Thrombectomy system,Thrombectomy system is an intraarterial thrombectomy removal device that can be re-inserted into the sheath to restore blood flow by removing blood clots in occluded vessels.
  Interventions: Device: Mechanical thrombectomy
- Intracranial thrombectomy stent :Solitaire FR Revascularization Device (Active Comparator): Subjects will be treated with Solitaire FR Revascularization Device ,the Device made by Micro Therapeutics Inc. DBA ev3 Neurovascular

INTERVENTIONS:
Device: Mechanical thrombectomy — Treatment of ischemic stroke patients with Mechanical thrombectomy
  Arms: Mechanical thrombectomy:Thrombectomy system

SUMMARY:
Through the implementation of prospective, multi-center, randomized, parallel controlled clinical studies to verify the safety and effectiveness of Hongyuan thrombolysis device system in the intravascular treatment of acute ischemic stroke. According to the requirements of the experiment, 200 subjects were selected and randomly divided into the experimental group and the control group 1:1. According to the information of the group, corresponding devices were used to receive endovascular therapy and the results were evaluated.

DETAILED DESCRIPTION:
Through the implementation of prospective, multi-center, randomized, parallel controlled clinical studies to verify the safety and effectiveness of Hongyuan thrombolysis device system in the intravascular treatment of acute ischemic stroke. According to the requirements of the trial, 200 subjects with acute ischemic stroke who met the inclusion criteria and did not meet any exclusion criteria were randomly divided into the test group and the control group at 1:1, and received endovascular therapy with corresponding instruments according to the information of the group and evaluated the results

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85
2. Within 8 hours of the onset of stroke symptoms
3. There are clinical signs and symptoms consistent with acute ischemic stroke
4. Imaging examination excluded intracranial hemorrhage, and there were no imaging changes of early large cerebral infarction (large infarction was defined as the aspect score of CT or DWI image < 6, infarct volume ≥70ml or infarct area > 1/3MCA)
5. Patients with imaging evidence of stroke caused by occlusion of the internal carotid artery (intracranial segment) or the M1/M2 segment of the middle cerebral artery or the A1/A2 segment of the anterior cerebral artery without clear contraindications
6. 6 points ≤NIHSS score < 30 points
7. Informed consent is signed by the patient or her legal guardian

Exclusion Criteria:

1. Known allergies to heparin, narcotic drugs, contrast agents, and/or antiplatelet medications such as aspirin and clopidogrel
2. mRS ≥ 2 before stroke
3. Pregnant Or Lactating Women
4. Hemorrhagic cerebrovascular history within 3 months
5. Refractory hypertension that cannot be controlled by medication (systolic blood pressure ≥185mmHg, or diastolic blood pressure ≥110mmHg)
6. Bleeding prone predisposition with severe coagulopathy, such as INR > 3.0 or platelet count < 40x10∧9/L
7. Blood glucose at screening was < 2.8mmol/L or > 22 mmol/L
8. Patients with any of the following exclusion criteria were not eligible to participate in this study

   * Preoperative CT or MRI showed bleeding symptoms
   * CT or MRI shows intracranial mass or intracranial tumor requiring surgical treatment
   * Angiography revealed carotid dissection or extracranial occlusion or arteritis of the carotid artery
   * Angiography revealed simultaneous acute obstruction of both carotid systems
9. Participate in other drug or device clinical trials within 28 days prior to screening visit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Immediate postoperative target vessel recanalization (mTICI≥2b) rate | Immediately after surgery
  According to 《the recommendations of the Chinese Guidelines for Stroke Prevention and Treatment》 , the therapeutic goal of mechanical thrombectomy is to achieve reperfusion of mTICI≥2b, so as to achieve the best possible functional outcome for patients. Therefore, we selected immediate postoperative target vessel recanalization (mTICI≥2b) rate as the primary efficacy endpoint.

SECONDARY OUTCOMES:
The time from puncture to recanalization | immediately after surgery
  The time from onset to recanalization will affect the prognosis of patients, and shorter recanalization time will bring better prognostic effect. Therefore, we chose the time from puncture to recanalization to compare the opening efficiency of the two groups of instruments.
The number of thrombectomy | immediately after surgery
  The number of thrombectomy will affect the rate of vascular opening and the mortality of subjects, so we selected the number of thrombectomy as indicators to evaluate the efficiency of the opening of the instrument.
the rate of successful vascular recirculation after the first thrombectomy | immediately after surgery
  The number of thrombectomy will affect the rate of vascular opening and the mortality of subjects, so we selected the rate of successful vascular recirculation after the first thrombectomy as indicators to evaluate the efficiency of the opening of the instrument.
NIHSS Score | 24hours and 7days after surgery
  The Assessment of Neurological Deficits (NIHSS score) is a well-established and widely accepted scale for evaluating neurological deficits in stroke patients. Neurological function evaluation (NIHSS score) at one day after endovascular therapy is helpful to predict clinical outcome at 90 days after surgery. A score of 3 is usually considered as the limit. A score of 3 or less indicates a mild stroke, a score of 3-10 is a moderate stroke, and a score of more than 10 is a severe stroke.
Proportion of patients with an mRS Score of 0-2 at 90 days after surgery | 3 mouths after surgery
  MRS Score, also known as modified Rankin score scale, is a scale used to evaluate the recovery state of neurological function in stroke patients. There are seven levels, level 0: completely asymptomatic. Level 1: Despite symptoms, the patient has no apparent disability and can perform all regular work and activities. Level 2: Mildly disabled, unable to perform all work and activities, but able to handle personal matters without assistance from others. Level 3: moderately disabled, requiring assistance, to walking without assistance. Level 4: Severely disabled, unable to walk without assistance, unable to care for their own needs. Level 5: Severely disabled, bedridden, incontinent, in need of constant care, and in need of multiple round-the-clock attention. Level 6: Dead .The proportion of subjects with mRS Score of 0-2 at 90 days after surgery was selected as the basis for judging the prognosis of subjects.
Performance evaluation of the device | immediately after surgery
  Device performance evaluation can help to evaluate the maneuverability of research devices in clinical application.Including the ability of the instrument to reach the lesion, the ability of the instrument to release and deploy smoothly, and the difficulty of the instrument to withdraw

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Xiangyang First People's Hospital, Xiangyang, Hubei
  - The first people's hospital of changzhou, Changzhou, Jiangsu
  - Zhangjiagang First People's Hospital, Suzhou, Jiangsu
  - The Second People's Hospital of Wuxi, Wuxi, Jiangsu
  - The affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Xianyang Hospital of Yan 'an University, Xianyang, Shanxi
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jiaxing Second Hospital, Jiaxing, Zhejiang
  - Lishui Municipal Central Hospital, Lishui, Zhejiang

IPD SHARING:
Plan to Share IPD: No